CLINICAL TRIAL: NCT06785571
Title: The Evaluation of the Effectiveness and Safety of Nalbuphine Hydrochloride Injection for Analgesia in ICU Patients: A Multicenter, Randomized, Single-blinded, Parallel, Two-step Trial
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Collaborators: Yichang Humanwell Pharmaceutical Co., Ltd., China (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-0407
Record Dates: First submitted 2025-01-09; First posted 2025-01-21 (Actual); Last update posted 2025-01-21 (Actual); Status verified 2024-10

CONDITIONS: Respiratory Insufficiency
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Nalbuphine; Hydromorphone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- lower loading dose of Nalbuphine hydrochloride for step 1 (Experimental): Nalbuphine hydrochloride injection, a loading dose of 4 mg administered in 30 ±10 seconds, followed by a maintenance dose of 2.0mg/h (a recommended maintenance dose range of 1.0~5.0mg/h)
  Interventions: Drug: Nalbuphine hydrochloride injection
- higher loading dose of Nalbuphine hydrochloride for step 1 (Experimental): Nalbuphine hydrochloride injection, a loading dose of 6 mg administered in 30 ±10 seconds, followed by a maintenance dose of 2.0mg/h (a recommended maintenance dose range of 1.0~5.0mg/h)
  Interventions: Drug: Nalbuphine hydrochloride injection
- Hydromorphone hydrochloride injection for step 1 (Active Comparator): Hydromorphone hydrochloride injection: a maintenance dose of 0.5mg/h (a recommended maintenance dose range of 0.5~3.0mg/h)
  Interventions: Drug: Hydromorphone hydrochloride injection
- The optimal loading of Nalbuphine hydrochloride injection for step 2 (Experimental): Nalbuphine hydrochloride injection: a loading dose determined after step 1 administered in 30 ±10 seconds, followed by a maintenance dose of 2.0mg/h (a recommended maintenance dose range of 1.0~5.0mg/h)
  Interventions: Drug: Nalbuphine hydrochloride injection
- Hydromorphone hydrochloride injection for step 2 (Active Comparator): Hydromorphone hydrochloride injection: a maintenance dose of 0.5mg/h (a recommended maintenance dose range of 0.5~3.0mg/h)
  Interventions: Drug: Hydromorphone hydrochloride injection

INTERVENTIONS:
Drug: Nalbuphine hydrochloride injection — a loading dose of Nalbuphine hydrochloride injection administered in 30 ±10 seconds, followed by a maintenance dose of 2.0mg/h (a recommended maintenance dose range of 1.0~5.0mg/h)
  Arms: The optimal loading of Nalbuphine hydrochloride injection for step 2; higher loading dose of Nalbuphine hydrochloride for step 1; lower loading dose of Nalbuphine hydrochloride for step 1
Drug: Hydromorphone hydrochloride injection — A maintenance dose of 0.5mg/h (a recommended maintenance dose range of 0.5~3.0mg/h)
  Arms: Hydromorphone hydrochloride injection for step 1; Hydromorphone hydrochloride injection for step 2

SUMMARY:
The analgesic effect of nalbuphine hydrochloride injection will be evaluated in a multicenter, randomized, single-blind, parallel, positive-controlled approach in two steps: step 1, to explore the optimal dosage of nalbuphine hydrochloride injection with 2 experimental arms and 1 positive control and step 2, to evaluate the effectiveness and safety of nalbuphine hydrochloride injection in mechanically ventilated ICU patients at a dosage determined in step 1 with the same positive control.

ELIGIBILITY:
Inclusion Criteria:

1. ICU patients who are intubated are expected to require mechanical ventilation for more than 6h
2. patients or their guardians have a full understanding of the purpose and significance of this trial, and voluntarily participate in this clinical trial and sign an informed consent form

Exclusion Criteria:

1. Allergy or unsuitability to any composition of study drugs or propofol
2. Living expectancy of less than 48 hours
3. Neurological disorder and any other condition interfering with sedation assessment
4. Gastrointestinal obstruction
5. Asthmatic
6. Abdominal compartment syndrome
7. Serious hepatic dysfunction (CTP 10-15)
8. Acute kidney injury (KDIGO stage 2 or 3) or Chronic kidney disease with glomerular filtration rate (GFR) < 29 ml/min/1.73m2
9. Circulatory instability (the need for a continuous infusion of norepinephrine at ≥0.5 ug/kg/min to maintain proper blood pressure)
10. Need deep sedation or paralytics
11. Anticipation to receive operations (including tracheotomy)
12. Abuse of controlled substances or alcohol
13. Pregnancy, lactation, or an intention of gestation in 6 months
14. Inclusion in another interventional trial in the past 30 days
15. Other conditions deemed unsuitable to be included

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2023-08-30 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
The analgesic success rate | Within 24 hours while receiving the study drug
  The analgesic success is determined as 1) no use of rescue analgesic medication and 2) at least 70% of the time with CPOT ≤ 2 points

SECONDARY OUTCOMES:
The percentage of time with light sedation duration | Within 24 hours while receiving the study drug
  Light sedation duration is defined as subjects with CPOT ≤ 2 points and -2 points ≤ RASS ≤ 1
The amout of propfol used | Within 24 hours while receiving the study drug
  The amout of propfol used
Successful extubation | Within 24 hours while receiving the study drug
  Successful extubated without reintubation

OTHER OUTCOMES:
Cmax | Within 24 hours while receiving the study drug
  peak plasma concentration
The area under the plasma drug concentration-time curve | Within 24 hours while receiving the study drug
  The area under the plasma drug concentration-time curve (AUC)
t1/2 | Within 24 hours while receiving the study drug
  half-life

CONTACTS AND LOCATIONS:
Locations (1):
- Wuhan Union Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No